CLINICAL TRIAL: NCT05676190
Title: Treatment of Colorectal Cancer With Autologous Cytokine Induced Killer Cells (CIK)
Brief Title: Clinical Study on the Efficacy of Autologous Cell Factor Induced Killer Cells in the Treatment of Colorectal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ShiCang Yu (Other)
Responsible Party: Sponsor-Investigator, ShiCang Yu, chief physician, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zsyx2
Record Dates: First submitted 2022-12-08; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer
Keywords: Autologous cytokine induced killer cells
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CIK combined with chemotherapy group (Experimental): Combination of CIK cells and chemotherapy
  Interventions: Combination Product: CIK combined with chemotherapy group
- CIK combined immunotherapy group (Experimental): Combination of CIK cells and immunotherapy
  Interventions: Combination Product: CIK combined immunotherapy group
- CIK combined targeted therapy group (Experimental): Combination of CIK cells and targeted therapy
  Interventions: Combination Product: CIK combined targeted therapy group
- CIK in combination with other therapies (Experimental): CIK in combination with any two or three of these (i.e., chemotherapy, immunotherapy, and targeted therapy) treatments
  Interventions: Combination Product: CIK in combination with other therapies

INTERVENTIONS:
Combination Product: CIK combined with chemotherapy group — Combination of chemotherapy and autologous cytokine induced killer cells
  Arms: CIK combined with chemotherapy group
Combination Product: CIK combined immunotherapy group — Combination of immunotherapy and autologous cytokine induced killer cells
  Arms: CIK combined immunotherapy group
Combination Product: CIK combined targeted therapy group — Combination of targeted therapy and autologous cytokine induced killer cells
  Arms: CIK combined targeted therapy group
Combination Product: CIK in combination with other therapies — CIK combined with any two or three of them (i.e. chemotherapy, immunotherapy and targeted therapy)
  Arms: CIK in combination with other therapies

SUMMARY:
This project plans to use CIK combined with chemotherapy, immunotherapy and targeted therapy to treat CRC patients, so as to explore the effectiveness of CIK treatment and the CRC subtypes more suitable for CIK treatment, thereby improving the survival rate and quality of life of CRC patients.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a malignant tumor that seriously threatens human health, and according to the international agency for research on cancer (IARC) data, in 2018, the number of new cases of CRC totalled more than 1.8 million and the number of deaths totalled more than 88million, making it the third most common cancer worldwide [1]. In recent years, with the development of economic level in China, changes in lifestyle and dietary structure, the incidence and mortality of CRC have shown a continuous increasing trend, and it is ranked 5th in all malignant tumors. According to statistics, at present, our country has 376000 new CRC cases and 191000 deaths annually, and the whole face extremely serious challenges.

Patients with advanced CRC have a more complicated disease, and the 5-year survival rate is even less than 5%. A single therapeutic means cannot achieve the desired therapeutic effect, and often multiple therapeutic modalities are used for intervention, including surgery, radiotherapy, chemotherapy, interventional minimally invasive treatment, immunotherapy and molecular targeting, etc. Because of the potential efficacy of CIK treatment in controlling tumor growth and prolonging patient survival, but there are still few clinical studies about CIK combined with other treatment modalities, this protocol is intended to use CIK combined with chemotherapy, immune and targeted therapy in CRC patients, in order to explore the effectiveness of CIK treatment and more suitable CRC subtypes for CIK treatment, and then improve the survival rate and quality of life of CRC patients.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-70 years;

  * Patients diagnosed with colorectal cancer, TNM stage III-IV;

    * Had at least one extracranially measurable lesion by recist1.1 criteria; ④ Patients who had failed at least one or two prior lines of standard therapy or relapsed, or who were intolerant to or voluntarily abandoned one or two prior lines of standard therapy; ⑤ Expected survival ≥ 90 days;

      * The major organs function normally; ⑦ The subject voluntarily joined this study, signed the informed consent, complied well and cooperated with the follow-up.

Exclusion Criteria:

* Had participated in other clinical trialists of drugs within 4 weeks before the start of the study;

  * Those who had hypertension that was inadequately controlled with a single antihypertensive agent (systolic blood pressure > 140 mmHg and diastolic blood pressure > 90 mmHg, as judged by the investigator), had myocardial ischemia or myocardial infarction of grade I or higher, arrhythmia of grade I and higher (including QT interval ≥ 440 MS), or cardiac dysfunction;

    * Those with a history of substance abuse who are unable to abstain or who have a history of mental disorders;

      * Presence of fungal, bacterial, viral, or other infections that are not controllable or require antibiotic therapy;

        * For subjects with prior chemotherapy use, ≥ grade 2 hematologic toxicity, or ≥ grade 3 nonhematologic toxicity according to nci-ctcae 5.0 criteria at enrollment; ⑥ Known presence of a history of HIV, or hepatitis B (HBsAg positive) or hepatitis C virus (anti HCV positive) nucleic acid test positive;

          * Presence of any indwelling catheter or drain (eg, biliary drain or pleural / peritoneal / pericardial catheter). Use of a dedicated central venous catheter was permitted (colostomy for patients with bowel cancer, percutaneous nephrostomy tube, indwelling Frey catheter, considered by the investigator for implications); ⑧ Presence of brain metastases, presence of a history or disease of the CNS such as seizure disorders, cerebral ischemia / hemorrhage, dementia, cerebellar disease, or any autoimmune disease involving the CNS;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-09 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) | up to 5 years
  Disease control rate of colorectal cancer
objective response rate (ORR) | up to 5 years
  objective response rate of colorectal cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Southwest Hospital, Army Medical University (Third Military Medical University), Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gammaitoni L, Giraudo L, Macagno M, Leuci V, Mesiano G, Rotolo R, Sassi F, Sanlorenzo M, Zaccagna A, Pisacane A, Senetta R, Cangemi M, Cattaneo G, Martin V, Coha V, Gallo S, Pignochino Y, Sapino A, Grignani G, Carnevale-Schianca F, Aglietta M, Sangiolo D. Cytokine-Induced Killer Cells Kill Chemo-surviving Melanoma Cancer Stem Cells. Clin Cancer Res. 2017 May 1;23(9):2277-2288. doi: 10.1158/1078-0432.CCR-16-1524. Epub 2016 Nov 4. PMID 27815354
- [Result] Garofano F, Gonzalez-Carmona MA, Skowasch D, Schmidt-Wolf R, Abramian A, Hauser S, Strassburg CP, Schmidt-Wolf IGH. Clinical Trials with Combination of Cytokine-Induced Killer Cells and Dendritic Cells for Cancer Therapy. Int J Mol Sci. 2019 Sep 3;20(17):4307. doi: 10.3390/ijms20174307. PMID 31484350
- [Result] Dienstmann R, Mason MJ, Sinicrope FA, Phipps AI, Tejpar S, Nesbakken A, Danielsen SA, Sveen A, Buchanan DD, Clendenning M, Rosty C, Bot B, Alberts SR, Milburn Jessup J, Lothe RA, Delorenzi M, Newcomb PA, Sargent D, Guinney J. Prediction of overall survival in stage II and III colon cancer beyond TNM system: a retrospective, pooled biomarker study. Ann Oncol. 2017 May 1;28(5):1023-1031. doi: 10.1093/annonc/mdx052. PMID 28453697